CLINICAL TRIAL: NCT04338893
Title: ROSA Total Knee Post Market Study: a Prospective, Multicenter EMEA Post Market Clinical Follow up of the ROSA Knee System
Brief Title: ROSA Total Knee Post Market Study EMEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CME2019-24K
Record Dates: First submitted 2020-01-24; First posted 2020-04-08 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Knee Pain; Chronic Osteoarthritis; Avascular Necrosis of the Femoral Condyle; Moderate Varus, Valgus or Flexion Deformities; Rheumatoid Arthritis
MeSH Terms: conditions — Genu Valgum; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSA Total Knee Robotic Instrumentation (Active Comparator): Total knee arthroplasty performed with ROSA Total Knee Robotic instrumentation
  Interventions: Procedure: Device: Persona Total Knee; Procedure: Device: NexGen Total Knee; Procedure: Device: Vanguard Total Knee
- Conventional TKA Instrumentation (Active Comparator): Total knee arthroplasty performed with conventional instrumentation
  Interventions: Procedure: Device: Persona Total Knee; Procedure: Device: NexGen Total Knee; Procedure: Device: Vanguard Total Knee

INTERVENTIONS:
Procedure: Device: Persona Total Knee — The choice of intervention is defined by surgeons standard use of device 'Persona' in their standard of care practice
Procedure: Device: NexGen Total Knee — The choice of intervention is defined by surgeons standard use of device 'Nexgen' in their standard of care practice
Procedure: Device: Vanguard Total Knee — The choice of intervention is defined by surgeons standard use of device 'Vanguard' in their standard of care practice

SUMMARY:
This is a prospective, multicenter clinical study designed to facilitate the collection and evaluation of surgical workflow efficiency, patient pain and function outcome and adverse events data. This study might include Persona, Nexgen and Vanguard product families using the ROSA Total Knee Robotic system or conventional instrumentation. The primary objective is to evaluate the accuracy of implant alignment for ROSA Total Knee robotic instrumentation compared to conventional instrumentation.

DETAILED DESCRIPTION:
The main purpose of this study is to collect and compare clinical outcomes data using the commercially available ROSA Total Knee robotic instrumentation and conventional instrumentation. This will be achieved by assessing: planned vs actual component positioning, operative workflow efficiency, patient safety based on incidence and frequency of adverse events, clinical performance measured by overall pain and function, health-related quality of life data and radiographic parameters.

The primary endpoint will report on the accuracy of implant alignment for ROSA Total Knee robotic instrumentation compared to conventional and the secondary endpoints will record surgery time points and evaluate the change of clinical outcomes scores between baseline and post operative follow up for performance and clinical benefits

ELIGIBILITY:
Inclusion/Exclusion criteria Inclusion criteria:

* Patient is a minimum of 18 years of age
* Independent of study participation, patient is a candidate for commercially available Persona, NexGen, or Vanguard knee components implanted in accordance with product labeling
* Patient has participated in this study-related Informed Consent Process
* Patient is willing and able to provide written Informed Consent by signing and dating the EC approved Informed Consent form
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations

Exclusion criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Patient has underwent contralateral UKA or TKA within the last 18 months
* Hip pathology with significant bone loss (e.g. avascular necrosis of the femoral head with collapse, severe dysplasia of the femoral head or the acetabulum)
* Hip pathology severely limiting range of motion (e.g. arthrodesis, severe contractures, chronic severe dislocation)
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (6):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Germany (2):
  - Herzogin Elisabeth Hospital, Braunschweig
  - Evangelisches Waldkrankenhaus Spandau, Spandau
- The Research Fund of Hadassah Medical Organization, Jerusalem, Israel
- San Giuseppe Hospital, Arezzo, Italy
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients not assigned to any group: 27 screen failures, 1 cancelled operation, 3 recorded as lost to follow-up for other reasons
Groups:
- Robotic: Total knee arthroplasty performed with ROSA Total Knee Robotic instrumentation
- Conventional: Total knee arthroplasty performed with conventional instrumentation
Period: Overall Study
Arm/Group | Robotic | Conventional
Started | 120 | 101
Completed | 85 | 75
Not Completed | 35 | 26
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Death | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 23 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic | Conventional | Total
Number analyzed (Participants) | 120 | 101 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (7.9) | 70.4 (8.7) | 70.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 66 | 141
  Male | 45 | 35 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Alignment Accuracy
Description: Evaluate the accuracy of implant component alignment for ROSA Total Knee robotic instrumentation compared to conventional instrumentation, by measuring femoral rotation in the axial plane using pre op and post op CT assessments.
Time Frame: Pre-operative, 3 months
Population: CT scans were taken from participants enrolled in this patients sub-cohort; however, following longer study duration and fewer enrolled patients than originally planned, the scans analysis was not performed, as the reduced sample size limited interpretability, resources were reallocated, and the research question was no longer considered novel.
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Operative Workflow Efficiency
Description: Measure operative workflow efficiency by recording following time points during surgery: Patient in -and out time, incision - and incision closed time
Time Frame: Intraoperative
Population: Information not collected for 2 conventional patients
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 99
minutes
  Time from patient in to patient out | 161.6 (30.9) | 138.8 (27.9)
  Time from incision cut to incision closed | 91.5 (21.1) | 77.5 (20.3)

3. Secondary Outcome: Oxford Knee Score (OKS)
Description: The OKS is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following TKA. The OKS consists of twelve questions covering function and pain associated with the knee. To calculate the total score, each question is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27
Time Frame: Pre-operative, 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
score on a scale
  Pre-operative: number analyzed (Participants) | 115 | 96
  Pre-operative | 21.5 (7.5) | 20.6 (6.8)
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks | 30.5 (7.1) | 29.0 (7.8)
  3 months: number analyzed (Participants) | 104 | 88
  3 months | 36.3 (8.0) | 35.0 (9.6)
  1 year: number analyzed (Participants) | 83 | 74
  1 year | 38.5 (8.9) | 38.2 (9.2)

4. Secondary Outcome: EuroQol 5D (EQ-5D) - Score
Description: The EQ-5D is a standardized instrument widely used to measure health status, and it is a self-reported assessment about the patient's quality of life. The questionnaire includes 5 questions referring to mobility, self-care, daily/usual activities, pain/discomfort and anxiety/depression. For EQ-5D-5L, each question can be answered in five ways, indicating no, slight, moderate, severe or extreme pain. In the derived EQ-5D-5L score, the highest score is 1 and the lowest score is -0.573; negative numbers correspond to a self-assessed health state worse than being dead.
Time Frame: Pre-operative, 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
score on a scale
  Pre-operative: number analyzed (Participants) | 116 | 96
  Pre-operative | 0.371 (0.336) | 0.388 (0.303)
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks | 0.717 (0.204) | 0.691 (0.232)
  3 months: number analyzed (Participants) | 104 | 88
  3 months | 0.816 (0.160) | 0.762 (0.266)
  1 year: number analyzed (Participants) | 84 | 74
  1 year | 0.865 (0.179) | 0.817 (0.238)

5. Secondary Outcome: EuroQol 5D (EQ-5D) VAS Scale
Description: The EQ-5D is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The VAS is a vertical scale ranging from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her self-rated health.
Time Frame: Pre-operative, 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
score on a scale
  Pre-operative: number analyzed (Participants) | 119 | 98
  Pre-operative | 64.8 (18.0) | 64.6 (20.0)
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks | 73.8 (15.1) | 73.9 (15.6)
  3 months: number analyzed (Participants) | 104 | 88
  3 months | 78.6 (15.4) | 78.1 (14.7)
  1 year: number analyzed (Participants) | 83 | 74
  1 year | 76.1 (18.8) | 78.6 (17.7)

6. Secondary Outcome: NRS (Numeric Rating Scale) Pain
Description: The NRS Pain is an outcome measure of pain intensity in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Scores range from 0-10 points, with 0 representing "no pain" to 10 representing "worst imaginable pain".
Time Frame: Pre-operative, 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
score on a scale
  Pre-operative | 7.2 (2.0) | 7.5 (1.5)
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks | 3.4 (2.0) | 3.2 (2.1)
  3 months: number analyzed (Participants) | 104 | 88
  3 months | 2.3 (2.2) | 2.3 (2.1)
  1 year: number analyzed (Participants) | 84 | 73
  1 year | 1.5 (2.0) | 1.7 (1.9)

7. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The FJS-12 is a patient-reported outcome questionnaire that was developed to specifically assess the patient's level of awareness of having a joint prosthesis during daily activities. The FJS consists of twelve questions covering function and pain associated with the knee. For each question, there is a choice of five answers between never (0), almost never (1), seldom (2), sometimes (3) and mostly (4). All scores are summed up and divided by the number of completed items. This value is then multiplied by 25 and thereafter subtracted from 100. An outcome score of 100 (highest possible score) indicates the lowest level of awareness of having a joint prosthesis, while a total score of 0 indicates the highest level of awareness of having a joint prosthesis.
Time Frame: Pre-operative, 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
score on a scale
  Pre-operative: number analyzed (Participants) | 116 | 96
  Pre-operative | 21.3 (14.5) | 17.6 (13.1)
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks | 42.4 (22.5) | 37.1 (22.1)
  3 months: number analyzed (Participants) | 103 | 88
  3 months | 60.5 (24.6) | 55.3 (26.2)
  1 year: number analyzed (Participants) | 83 | 73
  1 year | 67.4 (25.2) | 64.7 (27.2)

8. Secondary Outcome: Patient Satisfaction - Question 1
Description: Patients were asked to answer the following question: "How satisfied are you with the results of your surgery?" by selecting from the answers: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied.
Time Frame: 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
Participants
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks: Very satisfied | 54 | 49
  6 weeks: Somewhat satisfied | 42 | 29
  6 weeks: Somewhat dissatisfied | 8 | 10
  6 weeks: Very dissatisfied | 2 | 1
  3 months: number analyzed (Participants) | 104 | 88
  3 months: Very satisfied | 62 | 48
  3 months: Somewhat satisfied | 35 | 33
  3 months: Somewhat dissatisfied | 6 | 4
  3 months: Very dissatisfied | 1 | 3
  1 year: number analyzed (Participants) | 84 | 74
  1 year: Very satisfied | 50 | 44
  1 year: Somewhat satisfied | 31 | 25
  1 year: Somewhat dissatisfied | 3 | 4
  1 year: Very dissatisfied | 0 | 1

9. Secondary Outcome: Patient Satisfaction - Question 2
Description: Patients were asked to answer the following question: "How satisfied are you with the results of your surgery for improving your pain?" by selecting from the answers: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied.
Time Frame: 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
Participants
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks: Very satisified | 41 | 31
  6 weeks: Somewhat satisfied | 51 | 43
  6 weeks: Somewhat dissatisfied | 11 | 15
  6 weeks: Very dissatisfied | 3 | 0
  3 months: number analyzed (Participants) | 103 | 88
  3 months: Very satisified | 63 | 49
  3 months: Somewhat satisfied | 31 | 31
  3 months: Somewhat dissatisfied | 9 | 5
  3 months: Very dissatisfied | 0 | 3
  1 year: number analyzed (Participants) | 84 | 74
  1 year: Very satisified | 51 | 53
  1 year: Somewhat satisfied | 28 | 14
  1 year: Somewhat dissatisfied | 4 | 4
  1 year: Very dissatisfied | 1 | 3

10. Secondary Outcome: Patient Satisfaction - Question 3
Description: Patients were asked to answer the following question: "How satisfied are you with the results of your surgery for improving your ability to do home or yard work?" by selecting from the answers: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied.
Time Frame: 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
Participants
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks: Very satisified | 34 | 13
  6 weeks: Somewhat satisfied | 57 | 60
  6 weeks: Somewhat dissatisfied | 12 | 15
  6 weeks: Very dissatisfied | 3 | 1
  3 months: number analyzed (Participants) | 104 | 88
  3 months: Very satisified | 56 | 33
  3 months: Somewhat satisfied | 40 | 42
  3 months: Somewhat dissatisfied | 6 | 8
  3 months: Very dissatisfied | 2 | 5
  1 year: number analyzed (Participants) | 83 | 74
  1 year: Very satisified | 46 | 36
  1 year: Somewhat satisfied | 32 | 29
  1 year: Somewhat dissatisfied | 4 | 9
  1 year: Very dissatisfied | 1 | 0

11. Secondary Outcome: Patient Satisfaction - Question 4
Description: Patients were asked to answer the following question: "How satisfied are you with the results of your surgery for improving your ability to do recreational activities?" by selecting from the answers: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied.
Time Frame: 6 weeks, 3 months, 1 year
Population: Some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic | Conventional
Number analyzed (Participants) | 120 | 101
Participants
  6 weeks: number analyzed (Participants) | 106 | 89
  6 weeks: Very satisified | 34 | 17
  6 weeks: Somewhat satisfied | 54 | 52
  6 weeks: Somewhat dissatisfied | 14 | 16
  6 weeks: Very dissatisfied | 4 | 4
  3 months: number analyzed (Participants) | 104 | 88
  3 months: Very satisified | 55 | 37
  3 months: Somewhat satisfied | 37 | 36
  3 months: Somewhat dissatisfied | 10 | 10
  3 months: Very dissatisfied | 2 | 5
  1 year: number analyzed (Participants) | 82 | 74
  1 year: Very satisified | 45 | 43
  1 year: Somewhat satisfied | 33 | 22
  1 year: Somewhat dissatisfied | 3 | 9
  1 year: Very dissatisfied | 1 | 0

ADVERSE EVENTS:
Time Frame: From study start up to 1 year post-operatively
Description: Adverse events have been documented continuously by checking with the study patients at every follow-up visit.
Arm/Group | Robotic | Conventional
All-Cause Mortality (participants affected / at risk) | 0/120 | 1/101
Serious Adverse Events (participants affected / at risk) | 19/120 | 13/101
Other Adverse Events (participants affected / at risk) | 21/120 | 21/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic (N=120) | Conventional (N=101)
Infection (knee) (Surgical and medical procedures) | 1 | 0 — Required revision surgery
Post-operative cement leftover (Surgical and medical procedures) | 1 | 0 — Required revision surgery
Robotic malfunction (Product Issues) | 1 | 0
Effusion/Swelling/Edema (Blood and lymphatic system disorders) | 2 | 2
Vastus Lateralis Querruptur (Musculoskeletal and connective tissue disorders) | 0 | 1
Stiffness/Limited ROM (Musculoskeletal and connective tissue disorders) | 1 | 3 — Required manipulation under anesthesia
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Wound complication (Skin and subcutaneous tissue disorders) | 1 | 1
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Coronary heart disease (Cardiac disorders) | 1 | 0
Cardiac catheterization (Surgical and medical procedures) | 1 | 1
Shoulder replacement (Surgical and medical procedures) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Kidney Failure (Renal and urinary disorders) | 1 | 0
Cholecystitis (Surgical and medical procedures) | 1 | 0
Contralateral Knee Replacement (Surgical and medical procedures) | 2 | 2
Ureteral stenosis (Surgical and medical procedures) | 1 | 0
Nephrostomy (Surgical and medical procedures) | 1 | 0
Post-operative encephalopathy (Nervous system disorders) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 1 | 0
Discectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic (N=120) | Conventional (N=101)
Restricted Mobility Patella / Abnormal Patellar Tracking (Musculoskeletal and connective tissue disorders) | 6 | 6
Stiffness/Limited ROM (Musculoskeletal and connective tissue disorders) | 2 | 1
Effusion/Swelling/Edema (Vascular disorders) | 2 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dental-related problems (Musculoskeletal and connective tissue disorders) | 2 | 3
Covid infection (Infections and infestations) | 5 | 5
Tachycardia (Cardiac disorders) | 1 | 1
Heart surgery (Surgical and medical procedures) | 1 | 1
Eye surgery (Surgical and medical procedures) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT04338893/Prot_SAP_000.pdf